CLINICAL TRIAL: NCT02043860
Title: BMT-02: A Phase I Trial of Total Marrow Irradiation in Addition to High Dose Melphalan Conditioning Prior to Autologous Transplant for Multiple Myeloma Following Initial Induction Therapy
Brief Title: Total Marrow Irradiation With High Dose Melphalan Prior to Autologous Transplant for Multiple Myeloma
Acronym: BMT-02
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Pritesh Patel, MD, Faculty, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0202; 2013-0202 (Other: University of Illinois at Chicago)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; High Risk; Intermediate Risk; Symptomatic
MeSH Terms: conditions — Multiple Myeloma | interventions — Transplantation, Autologous; Melphalan; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Total Marrow Irradiation (Experimental): Escalating doses of total marrow irradiation (3Gy, 6Gy, 9Gy, or 12Gy) with standard high dose melphalan prior to autologous stem cell rescue.
  Interventions: Radiation: Total Marrow Irradiation; Procedure: Autologous Transplant; Drug: Melphalan; Drug: Filgrastim (G-CSF)

INTERVENTIONS:
Radiation: Total Marrow Irradiation — Subjects in this trial will receive total body irradiation (3Gy) per day for up to four days and as little as one day. Total IMT doses: 3Gy, 6Gy, 9Gy, or 12Gy.
Procedure: Autologous Transplant — Subjects will receive standard melphalan 200mg/m^2 (100mg/m^2 day-2 and day-1) conditioning with escalating doses of total marrow irradiation prior to autologous stem cell rescue.
Drug: Melphalan — Subjects will receive standard melphalan 200mg/m^2 (100mg/m^2 day-2 and day-1) conditioning therapy prior to transplant.
  Other Names: Alkeran ®
Drug: Filgrastim (G-CSF) — Subjects to begin GCSF 5 μg/kg/d SC or IV on Day 5 and continue until ANC > 1000/mm^3 over period of 3 days.
  Other Names: Neupogen®

SUMMARY:
In this phase I trial, patients with multiple myeloma will receive standard high dose melphalan with autologous stem cell rescue. In addition the pre-transplant conditioning will include targeted total marrow irradiation (TMI). This conventional 3+3 phase I trial will increase the dose of TMI until the maximum tolerated dose (MTD) is reached. Initial patients enrolled will receive the lowest possible dose of 3Gy. Maximum dose will be 12Gy.

DETAILED DESCRIPTION:
To establish the maximal tolerated dose of total marrow irradiation which can be added to high dose melphalan conditioning in patients with multiple myeloma undergoing autologous stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting criteria for symptomatic myeloma
2. Patients must be high or intermediate risk of disease progression as defined by having one of the following criteria: 2.1 ISS stage 2 or 3 disease 2.2 Abnormal metaphase cytogenetics 2.3 Presence of FISH abnormalities aside from hyperdiploidy
3. Patients who have received at least 2 cycles of systemic treatment of any kind in the preceding 12 months
4. Patient age 18-75 years at time of enrollment
5. Karnofsky performance status of ≥70
6. Cardiac function: LVEF >40%
7. Hepatic: Bilirubin <2x upper limit of normal and ALT and AST < 2.5x the upper limit of normal
8. Renal: Creatinine clearance of ≥30mL/min, estimated or calculated
9. Pulmonary: DLCO, FEV1, FVC >50% of predicted (after correction for hemoglobin)

Exclusion Criteria:

1. Patients with diagnosis of plasma cell leukemia
2. Patients with myeloma who have had any disease progression prior to enrollment
3. Patients with truly non secretory myeloma (patients with light chain disease are eligible)
4. Pregnant or breast-feeding
5. Uncontrolled viral, fungal or bacterial infection Note: Infection is permitted if there is evidence of response to medication. Eligibility of HIV infected patients will be determined on a case-by-case basis.
6. Patients who have undergone prior allograft or autologous transplant
7. Prior solid organ transplant
8. Patients receiving prior radiation to more than 20% of bone marrow containing areas

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2016-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pritesh Patel, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- UIC Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 ineligible
Groups:
- Total Marrow Irradiation: Escalating doses of total marrow irradiation (3Gy(gray), 6Gy, 9Gy, or 12Gy) with standard high dose melphalan prior to autologous stem cell rescue.
  Total Marrow Irradiation (TMI): Subjects in this trial will receive total body irradiation (3Gy) per day for up to four days and as little as one day. Total IMT doses: 3Gy, 6Gy, 9Gy, or 12Gy.
  Autologous Transplant: Subjects will receive standard melphalan 200mg/m^2 (100mg/m^2 day-2 and day-1) conditioning with escalating doses of total marrow irradiation prior to autologous stem cell rescue.
  Melphalan: Subjects will receive standard melphalan 200mg/m^2 (100mg/m^2 day-2 and day-1) conditioning therapy prior to transplant.
  Filgrastim (G-CSF): Subjects to begin GCSF 5 μg/kg/d SC or IV on Day 5 and continue until ANC > 1000/mm^3 over period of 3 days.
Period: Overall Study
Arm/Group | Total Marrow Irradiation
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Marrow Irradiation
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival No Results Due to 1 Subject Came Off Treatment Within 7 Days and 1 Subject Came Off Treatment Within 5 Days. Not Enough Data to Analyze
Description: To evaluate progression free survival (PFS) and in patients with multiple myeloma undergoing autologous stem cell transplant using the combination of high dose melphalan and total marrow irradiation.
Time Frame: Up to 1 year post-transplant.
Population: Data not collected
Groups:
- Cohort 1 TMI Dose 3Gy: Cohort 1 patients will receive standard high dose melphalan with autologous stem cell rescue. Plus TMI at a dose of 3Gy.
Arm/Group | Cohort 1 TMI Dose 3Gy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Cohort 1 TMI Dose 3Gy: This is a phase I trial. Patients will receive standard high dose melphalan with autologous stem cell rescue. In addition the pre-transplant conditioning will include targeted total marrow irradiation (TMI). The dose of TMI will increase until the maximum tolerated dose (MTD) is reached. 3 participants will be in each cohort beginning with the lowest possible dose of 3Gy to a maximum dose of 12Gy.
  All Cause Mortality Total 0/2 0%
  Serious Adverse Events Total 0/2 0%
  Adverse Events not including serious adverse events Total 2/2 100% Oral Mucositis 2/2 100% Diarrhea 2/2 100% Nausea 1/2 50% Non-productive cough 1/2 50% Rash to face and back 1/2 50% Throat pain 1/2 50% GI bleed 1/2 50%
Arm/Group | Cohort 1 TMI Dose 3Gy
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 TMI Dose 3Gy (N=2)
Mucositis (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
GI bleed (Gastrointestinal disorders) | 1 (1)
Throat pain (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rash to face and back (Skin and subcutaneous tissue disorders) | 1 (1)
Non-productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only 2 subjects received total marrow irradiation at 3Gy dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No